CLINICAL TRIAL: NCT02800798
Title: Correlation Between Preeclampsia and Positive for Obstructive Sleep Apnea Screening Test: STOPBANG Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Lisa Sangkum, Doctor, Ramathibodi Hospital
Other Study IDs: Ramathibodi
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive sleep apnea; Preeclampsia; Pregnancy; Stopbang
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pre-Eclampsia

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High risk for OSA: High risk OSA defines as Stop-bang score ≥ 3
  Interventions: Other: Preeclampsia positive
- Low risk for OSA: Low risk OSA defines as Stop-bang score < 3
  Interventions: Other: Preeclampsia positive

INTERVENTIONS:
Other: Preeclampsia positive
  Other Names: Preeclampsia negative

SUMMARY:
The purpose of this study is to find the correlation between high risk OSA (obstructive sleep apnea) patient, based on Stop-bang screening tool and preeclampsia

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) has been associated with preeclampsia and intrauterine growth retardation (IUGR).

Since the gold standard diagnosis of OSA is polysomnogram which is limited by cost and availability. Therefore, various screening tools were proposed in order to identify high risk OSA patient such as Stop-bang questionnaire.

From the previous study, Stop-bang showed a high predictive performance and the score equal or higher than 3 determines high risk for OSA.

ELIGIBILITY:
Inclusion Criteria:

- Pregnant women who were scheduled for cesarean delivery or admitted to the antepartum unit at Ramathibodi hospital

Exclusion Criteria:

* Age < 18 year old
* Previous diagnose OSA
* Patients who have used continuous positive airway pressure (CPAP) or bi-level positive airway pressure (Bi-PAP) fro OSA treatment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thai pregnant women who were scheduled for cesarean delivery or vaginal delivery at Ramathibodi hospital
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of pre-eclampsia between high and low risk of OSA patient based on Stop-bang screening test | 1 day

SECONDARY OUTCOMES:
prevalence of pre-eclampsia between high and low risk of OSA patient, based on Epworth sleepiness scale | 1 day
prevalence of pre-eclampsia between high and low risk of OSA patient, based on Berlin questionnaire | 1 day
prevalence of pre-eclampsia between high and low risk of OSA patient, based on American society check list | 1 day
The prevalence of maternal adverse event between high risk and low risk of OSA patient | 1 day
  Maternal adverse events include hypoxemia, arrythmia, perioperative myocardial infarction, heart failure
The prevalence of neonatal adverse event between high risk and low risk of OSA patient | 1 day
  Neonatal adverse events include IUGR, neonatal intensive care unit admission, low apgar score

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Pengo MF, Rossi GP, Steier J. Obstructive sleep apnea, gestational hypertension and preeclampsia: a review of the literature. Curr Opin Pulm Med. 2014 Nov;20(6):588-94. doi: 10.1097/MCP.0000000000000097. PMID 25250803
- [Background] Antony KM, Agrawal A, Arndt ME, Murphy AM, Alapat PM, Guntupalli KK, Aagaard KM. Association of adverse perinatal outcomes with screening measures of obstructive sleep apnea. J Perinatol. 2014 Jun;34(6):441-8. doi: 10.1038/jp.2014.25. Epub 2014 Mar 6. PMID 24603455